CLINICAL TRIAL: NCT03220854
Title: Phase 2 Clinical Trial of Stereotactic Radiotherapy (SRT) and PD-1 or PD-L1 Inhibiting Therapy for Treatment of Advanced Solid Tumors After Disease Control on PD-1 or PD-L1 Inhibiting Therapy
Brief Title: SBRT + PD-1/PDL-1 Inhibiting Therapy for Advanced Solid Tumors After Dz Control on PD-1/PDL-1 Tx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16-12436; P30CA016059 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Steriotactic Radiotherapy followed by a commercially available PD-1 or PD-L1 inhibitor drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- A: SBRT (body) irradiation only (Experimental): Patients will receive a standard treatment regimen of SRT (refer to Section 6.3). The term SRT encompasses all radiotherapy using a stereotactic setup, both stereotactic radiosurgery (SRS) for metastatic lesions in the brain and stereotactic body radiotherapy (SBRT) for SRT delivered to all other locations
  Interventions: Radiation: Stereotactic radiotherapy; Other: Biological: humanized anti-PD-1 monoclonal antibody; Other: Biological: humanized anti-PD-L1 monoclonal antibody
- B: Patients receiving SBRT and SRS (body and brain) irradiation (Experimental): Patients will receive a standard treatment regimen of SRT (refer to Section 6.3). The term SRT encompasses all radiotherapy using a stereotactic setup, both stereotactic radiosurgery (SRS) for metastatic lesions in the brain and stereotactic body radiotherapy (SBRT) for SRT delivered to all other locations
  Interventions: Radiation: Stereotactic radiotherapy; Other: Biological: humanized anti-PD-1 monoclonal antibody; Other: Biological: humanized anti-PD-L1 monoclonal antibody
- C: Patients receiving SRS (brain) irradiation only (Experimental): Patients will receive a standard treatment regimen of SRT (refer to Section 6.3). The term SRT encompasses all radiotherapy using a stereotactic setup, both stereotactic radiosurgery (SRS) for metastatic lesions in the brain and stereotactic body radiotherapy (SBRT) for SRT delivered to all other locations
  Interventions: Radiation: Stereotactic radiotherapy; Other: Biological: humanized anti-PD-1 monoclonal antibody; Other: Biological: humanized anti-PD-L1 monoclonal antibody

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Treatment will be planned to deliver a total of 18 to 60 Gy to the planning target volume (PTV) in 3 to 5 fractions over 1 to 2 weeks.
  Other Names: SRT
Other: Biological: humanized anti-PD-1 monoclonal antibody — Standard of Care - patient will continue to be given the same PD-1 inhibitor they were receiving prior to study registration
  Other Names: PD-1
Other: Biological: humanized anti-PD-L1 monoclonal antibody — Standard of Care - patient will continue to be given the same PD-L1 inhibitor they were receiving prior to study registration
  Other Names: PD-L1

SUMMARY:
The purpose of this study is to find out if having radiation therapy and continuing immunotherapy can improve the benefit of immunotherapy. There have been reports of patients who were treated with radiation therapy that not only caused the treated tumors to shrink or stop growing, but also resulted in tumors that had not been treated in other parts of the body to shrink or stop growing. This effect is thought to be brought about by cells in the body's immune system that become active as a result of the effects of radiation therapy. If radiation therapy can stimulate the immune system, it may be possible for immunotherapy to be helpful again in treating a cancer that the immunotherapy drug helped treat before. This study will also check if receiving immunotherapy at the end of radiation therapy has any effect on the side effects of radiation therapy or immunotherapy.

DETAILED DESCRIPTION:
Stereotactic radiotherapy (SRT) will be delivered in up to 10 treatment fractions over 1 to 2 weeks. Patients will continue to receive the same FDA-approved programmed death receptor-1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitor that they had been receiving at the time of disease progression through 52 weeks following completion of SRT.

Correlative blood samples will be collected at baseline, prior to the second SRT fraction, after the last SRT fraction (on the same day), and at 8, 24, and 52 weeks after the last SRT fraction. These samples will be used to determine the mechanistic immunologic effects of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-proven diagnosis of a solid tumor malignancy
* One of the following criteria must be met:
* Clinical or radiographic evidence of disease control (defined as best response of stable disease (SD) or partial response (PR) or combination of both for ≥ 16 weeks) without evidence of complete response (CR) or progression OR
* Clinical or radiographic evidence of disease progression during treatment with PD-1 or PD-L1 inhibiting therapy, following previous tumor response (CR, PR, or SD for ≥ 16 weeks) to PD-1 or PD-L1 inhibiting therapy, and, for patients who discontinued PD-1 or PD-L1 inhibiting therapy during response to therapy, disease progression must have occurred following at least 8 weeks of re-treatment with PD-1 or PD-L1 inhibiting therapy Note: Both the treating medical oncologist and radiation oncologist must be in agreement with determination of disease progression.
* Administration of a PD-1 or PD-L1 inhibitor within 60 days prior to study registration
* Determination by the treating radiation oncologist that the patient is a candidate for SRT (ie, radiation therapy with a stereotactic setup) Note: All brain metastases will receive stereotactic radiotherapy (SRT).
* The total number of tumors requiring SRT must be ≤ 5 Note: Regardless of the number of brain metastases that will be treated with SRT, the brain metastases will be considered to be one tumor.
* Measurable disease by RECIST v1.1 that will not undergo SRT and that is amenable to monitoring Note: all brain metastases will receive SRT. Therefore, a patient with brain metastases that will be treated with SRT must also have extracranial disease that will not undergo SRT and that is amenable to monitoring
* Determination by the treating medical oncologist that the patient is a candidate to continue the PD-1 or PD-L1 inhibiting therapy that had previously provided disease control
* Age ≥ 18 years
* Karnofsky Performance Status score of ≥ 60 %
* A woman of childbearing potential (WCBP), defined as a woman who is < 60 years of age and has not had a hysterectomy, must have a documented negative serum pregnancy test within 14 days prior to initiating study treatment
* Ability to understand and willingness to sign the consent form

Exclusion Criteria:

* Other anti-cancer therapy administered between the time of tumor response to PD-1 or PD-L1 therapy and time of study enrollment Note: Patients treated with a combination of PD-1 or PD-L1 inhibiting therapy and other immunotherapy are eligible; patients taking hormonal anti-cancer therapies or steroids for central nervous system (CNS) edema management that, in the opinion of the investigator, are appropriate to continue are eligible.
* Any prior PD-1/PD-L1 therapy-related AE that, in the opinion of the investigator, warrants exclusion from participation in this trial
* Administration of any investigational agent within 4 weeks prior to initiating study treatment
* Known active hepatitis B or C
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Urdaneta, M.D., Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants enrolled in Arm B.
Groups:
- A: Patients Receiving SBRT (Body) Irradiation Only; B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation; C: Patients Receiving SRS (Brain) Irradiation Only: Patients will receive a standard treatment regimen of SRT (refer to Section 6.3). The term SRT encompasses all radiotherapy using a stereotactic setup, both stereotactic radiosurgery (SRS) for metastatic lesions in the brain and stereotactic body radiotherapy (SBRT) for SRT delivered to all other locations
Period: Overall Study
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Started | 4 | 0 | 1
Completed | 4 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants enrolled on Arm B
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only | Total
Number analyzed (Participants) | 4 | 0 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 3 | 0 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 68 [59 to 71] |  | 67 [67 to 67] | 67.8 [59 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 0 | 2
  Male | 2 |  | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0 | 0
  Not Hispanic or Latino | 4 |  | 1 | 5
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 4 |  | 0 | 4
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Improved Disease Control
Description: 1. Number of patients with improved disease control at 24 weeks following RT [Time Frame: up to 24 weeks following RT] 1a. Number of participants with improved disease control (SD, PR or CR) at 24 weeks per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) 1b. For participants enrolled with brain metastases: number of participants with improved disease (SD, PR or CR) control at 24 weeks per per Response Assessment in Neuro-Oncology for Brain Metastases (RANO-BM)
Time Frame: Up to 24 weeks following SRT
Population: No participants enrolled in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | A: SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants
  1a: Number of participants with improved disease control: Complete Response | 0 | 0 | 0
  1a: Number of participants with improved disease control: Partial Response | 0 | 0 | 0
  1a: Number of participants with improved disease control: Stable Disease | 0 | 0 | 0
  1a: Number of participants with improved disease control: Progression at or before 24 Weeks | 2 | 0 | 1
  1a: Number of participants with improved disease control: Not Evaluable | 2 | 0 | 0
  1b: Participants enrolled with brain metastases number of participants with improved disease control: Complete Response | NA — Group A participants did not receive brain irradiation | 0 | 0
  1b: Participants enrolled with brain metastases number of participants with improved disease control: Partial Response | NA — Group A participants did not receive brain irradiation | 0 | 0
  1b: Participants enrolled with brain metastases number of participants with improved disease control: Stable Disease | NA — Group A participants did not receive brain irradiation | 0 | 1
  1b: Participants enrolled with brain metastases number of participants with improved disease control: Progression at or before 24 Weeks | NA — Group A participants did not receive brain irradiation | 0 | 0
  1b: Participants enrolled with brain metastases number of participants with improved disease control: Not Evaluable | NA — Group A participants did not receive brain irradiation | 0 | 0

2. Secondary Outcome: Number of Patients Alive and Free From Progression at 24 Weeks Following SRT Per Unidimensional Immune-related Response Criteria (irRC)
Description: Number of participants alive and without progression (irSD+irPR+irCR) at 24 weeks post-RT per unidimensional immune-related response criteria (irRC)
  1b. For participants enrolled with brain metastases: number of participants alive and without progression (SD+PR+CR) at 24 weeks post-RT per immune Response Assessment in Neuro-Oncology (iRANO)
Time Frame: Up to 24 weeks following SRT
Population: No participants were enrolled in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants
  1a. Number of participants alive and without progression: Progression Free Survival per irRC at 24 wks | 0 | 0 | 0
  1a. Number of participants alive and without progression: Progression per irRC at or before 24 Weeks | 1 | 0 | 1
  1a. Number of participants alive and without progression: Not Evaluable | 3 | 0 | 0
  1b.For participants enrolled with brain metastases: Progression Free Survival per irRC at 24 wks | NA — Group A participants did not receive brain irradiation | 0 | 1
  1b.For participants enrolled with brain metastases: Progression per irRC at or before 24 Weeks | NA — Group A participants did not receive brain irradiation | 0 | 0
  1b.For participants enrolled with brain metastases: Not Evaluable | NA — Group A participants did not receive brain irradiation | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment Response in Irradiated Tumor Sites
Description: Number of participants with treatment response in irradiated tumor sites at 24 weeks post-RT.
Time Frame: Up to 24 weeks following SRT
Population: No participants enrolled on Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants
  Complete Response at Irradiated Sites | 0 |  | 0
  Partial Response at Irradiated Sites | 0 |  | 1
  Stable Disease at Irradiated Sites | 0 |  | 0
  Not assessed at week 24 due to overall progression | 2 |  | 0
  Not Evaluable | 2 |  | 0

4. Secondary Outcome: Number of Participants With Treatment Response in Non-irradiated Tumor Sites
Description: Number of participants with treatment response in non-irradiated tumor sites at 24 weeks post-RT
Time Frame: Up to 24 weeks post-RT
Population: No participants enrolled on Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | A: SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants
  Complete Response at non-irradiated sites | 0 |  | 0
  Partial Response at non-irradiated sites | 0 |  | 0
  Stable Disease at non-irradiated sites | 0 |  | 0
  Progression at non-irradiated sites at or before 24 weeks | 2 |  | 1
  Not Evaluable | 2 |  | 0

5. Secondary Outcome: Number of Patients Alive
Description: Number of patients who are alive at 2 years after completion of SRT
Time Frame: 2 years following SRT
Population: No participants enrolled on Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants
  Number of participants meeting 2 year survival threshold | 2 | 0 | 1
  Number of participants not meeting 2 year survival threshold | 1 | 0 | 0
  Not evaluable | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Grade 3 or Greater Toxicity
Description: Number of participants with grade 3 or greater toxicity from the regimen through 8 weeks following RT
Time Frame: Through 8 weeks following SRT
Population: No participants enrolled in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Immune-related Toxicity From the Regimen
Description: Number participants with immune-related AEs (irAEs) that require both checkpoint-inhibitor discontinuation and initiation of steroids reported per CTCAE v5.0
Time Frame: Up to 2 years following RT
Population: No participants enrolled on Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants
  Participants with immune-related AEs (irAEs) | 1 |  | 0
  Participants with no immune related AE's (irAEs) | 2 |  | 1
  Not Evaluable | 1 |  | 0

8. Secondary Outcome: Radiobiological Signatures Associated With the Regimen
Description: Number participants with samples collected and number of participants with samples analyzed for immunologic effects of the regimen
Time Frame: Up to 52 weeks post SRT
Population: No participants enrolled on Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
Number analyzed (Participants) | 4 | 0 | 1
Participants
  Number of participants with samples collected | 3 |  | 1
  Number of participants with samples analyzed for immunologic effects of the regimen | 0 | 0 | 0
  Number of participants with no samples collected | 1 |  | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from the time of first SRT fraction and continued until 8 weeks following completion of SRT.
Description: There were no participants enrolled on Arm B.
Arm/Group | A: Patients Receiving SBRT (Body) Irradiation Only | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation | C: Patients Receiving SRS (Brain) Irradiation Only
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 3/4 | 0/0 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Patients Receiving SBRT (Body) Irradiation Only (N=4) | B: Patients Receiving SBRT and SRS (Body and Brain) Irradiation (N=0) | C: Patients Receiving SRS (Brain) Irradiation Only (N=1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Incomplete objectives due to early closure to accrual of trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03220854/Prot_SAP_000.pdf